CLINICAL TRIAL: NCT01195688
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (1-700 mg) of BI 638683 Powder in Bottle (PiB) in Healthy Male Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: Safety and Tolerability of BI 638683 After Single Rising Oral Doses in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1279.1; 2010-021187-15 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Healthy

ARMS (2):
- BI 638683 (Experimental): 1 single dose per subject as oral solution
  Interventions: Drug: BI 638683 or placebo
- Placebo solution (Placebo Comparator): 1 single dose per subject as oral solution
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: BI 638683 or placebo — oral doses given to 6 subjects per dose group
  Arms: BI 638683
Drug: Placebo solution — oral doses given to 2 subjects per dose group
  Arms: Placebo solution

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 638683 in healthy male volunteers following oral administration of single rising doses

ELIGIBILITY:
Inclusion criteria:

healthy male subjects

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety of BI 638683 will be assessed in a descriptive way. | up to 14 days post treatment
Tolerability of BI 638683 will be assessed in a descriptive way. | up to 14 days post treatment

SECONDARY OUTCOMES:
To assess pharmacodynamics of BI 638683. | up to 5 days post study drug administration
To assess pharmacokinetics of BI 638683. | up to 5 days post study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1279.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany